CLINICAL TRIAL: NCT01030861
Title: AntiCD3 Mab (Teplizumab) For Prevention of Diabetes In Relatives At-Risk for Type 1 Diabetes Mellitus
Brief Title: Teplizumab for Prevention of Type 1 Diabetes In Relatives "At-Risk"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Research Resources (NCRR) (NIH); Juvenile Diabetes Research Foundation (Other); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TrialNet - tep (IND); UC4DK106993 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Autoantibody Positive; Non-diabetic Relatives at Risk for Type 1 Diabetes; High Risk; Impaired Glucose Tolerance
Keywords: type 1 diabetes; pre-diabetic; autoantibody positive; at risk for type 1 diabetes; glucose intolerance; relatives of people with type 1 diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teplizumab (Active Comparator): Intravenous infusions of teplizumab given for 14 consecutive days. Each infusion takes about 30 minutes and is followed by a 2 hour observation period.
  Interventions: Drug: Teplizumab
- Placebo infusion (Placebo Comparator): Intravenous infusion of placebo (saline) will be given for 14 consecutive days. Infusions will take approximately 30 minutes and will be followed by a two hour observation period.
  Interventions: Drug: Placebo infusion

INTERVENTIONS:
Drug: Teplizumab — intravenous infusions
  Arms: teplizumab
Drug: Placebo infusion — Placebo for Teplizumab
  Arms: Placebo infusion

SUMMARY:
The study will determine whether the anti-CD3 monoclonal antibody, teplizumab, can help to prevent or delay the onset of type 1 diabetes (T1D) in relatives determined to be at very high risk for developing the disease. Teplizumab has been studied in new onset type 1 diabetes for testing of efficacy and safety in previous studies; other studies are currently in progress. The results of previous studies indicate that teplizumab reduces the loss of insulin production during the first year after diagnosis in individuals with type 1 diabetes. The purpose of this study is to determine if teplizumab can interdict the immune process that causes the destruction of insulin secreting beta cells in the pancreas during the "pre-diabetic" state and thereby prevent or delay the onset of type 1 diabetes.

DETAILED DESCRIPTION:
The study plans to enroll approximately 71 subjects between the ages of 8-45 years, over 2-3 years. The study is projected to last between 4-6 years, depending upon rate of enrollment and number of subjects who develop diabetes.

The main study objective is to determine whether intervention with teplizumab will prevent or delay the development of type 1 diabetes in high risk autoantibody positive non-diabetic relatives of individuals with T1D. Secondary outcomes are to include analyses of C-peptide and other measures from Oral Glucose Tolerance Testing (OGTT), safety, tolerability, and other mechanistic outcomes will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 8-45 years
* Have a relative with type 1 diabetes
* If first degree relative must be 8-45 years old (brother, sister, parent, offspring)
* If second degree relative must be between 8-20 years old (niece, nephew, aunt, uncle, grandchild, cousin)
* Abnormal glucose tolerance by OGTT confirmed with 7 weeks of baseline visit [fasting blood glucose greater than 110mg/dL or and less than 126 mg/dL OR 2 hour glucose greater or equal to 140 mg/dL and less than 200 mg/dL OR 30, 60, or 90 minute value on OGTT greater than or equal to 200 mg/dL]
* Presence of at least two confirmed diabetes autoantibodies

Exclusion Criteria:

* type 1 diabetes previously diagnosed or detected at screening [fasting glucose greater or equal to 126 mg/dL or 2 hour glucose greater or equal to 200 mg/dL]
* abnormalities in blood counts, liver enzymes, international normalised ratio (INR),
* positive purified protein derivative (PPD) test

  * vaccination with live virus within 6 weeks of randomization
* evidence of acute infection based on laboratory testing or clinical evidence
* serological evidence of past current or past HIV , hepatitis B, or hepatitis C infection
* Be currently pregnant or lactating
* Prior treatment with study drug
* Prior treatment with other monoclonal antibody in past one year

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (19):
- United States (17):
  - University of California in San Francisco, San Francisco, California
  - University of California-San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes/ University of Colorado, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Benaroya Research Institute, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Forschergruppe Diabetes, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository: https://repository.niddk.nih.gov/studies/tn10-anti-cd3-prevention/?query=trialnet%20Teplizumab
URL: https://repository.niddk.nih.gov/studies/tn10-anti-cd3-prevention/?query=trialnet%20Teplizumab

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Lledo-Delgado A, Preston-Hurlburt P, Currie S, Clark P, Linsley PS, Long SA, Liu C, Koroleva G, Martins AJ, Tsang JS, Herold KC. Teplizumab induces persistent changes in the antigen-specific repertoire in individuals at risk for type 1 diabetes. J Clin Invest. 2024 Aug 13;134(18):e177492. doi: 10.1172/JCI177492. PMID 39137044
- [Derived] Novograd J, Frishman WH. Teplizumab Therapy to Delay the Onset of Type 1 Diabetes. Cardiol Rev. 2024 Nov-Dec 01;32(6):572-576. doi: 10.1097/CRD.0000000000000563. Epub 2023 May 9. PMID 37158990
- [Derived] Leung SS, Borg DJ, McCarthy DA, Boursalian TE, Cracraft J, Zhuang A, Fotheringham AK, Flemming N, Watkins T, Miles JJ, Groop PH, Scheijen JL, Schalkwijk CG, Steptoe RJ, Radford KJ, Knip M, Forbes JM. Soluble RAGE Prevents Type 1 Diabetes Expanding Functional Regulatory T Cells. Diabetes. 2022 Sep 1;71(9):1994-2008. doi: 10.2337/db22-0177. PMID 35713929
- [Derived] Herold KC, Bundy BN, Long SA, Bluestone JA, DiMeglio LA, Dufort MJ, Gitelman SE, Gottlieb PA, Krischer JP, Linsley PS, Marks JB, Moore W, Moran A, Rodriguez H, Russell WE, Schatz D, Skyler JS, Tsalikian E, Wherrett DK, Ziegler AG, Greenbaum CJ; Type 1 Diabetes TrialNet Study Group. An Anti-CD3 Antibody, Teplizumab, in Relatives at Risk for Type 1 Diabetes. N Engl J Med. 2019 Aug 15;381(7):603-613. doi: 10.1056/NEJMoa1902226. Epub 2019 Jun 9. PMID 31180194
- See also: Type 1 Diabetes TrialNet — https://www.diabetestrialnet.org/publicationsdatabase/Article

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teplizumab | Placebo Infusion
Started | 44 | 32
Completed | 44 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teplizumab | Placebo Infusion | Total
Number analyzed (Participants) | 44 | 32 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [8.5 to 49.5] | 13 [8.6 to 45.0] | 13.9 [11.5 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 25 | 17 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 43 | 31 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 30 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Relationship to person with type 1 diabetes [Count of Participants; unit: Participants]
  Sibling(s) | 24 | 16 | 40
  Identical twin | 4 | 0 | 4
  Offspring | 6 | 6 | 12
  Parent | 6 | 3 | 9
  Sibling and another first degree relative | 2 | 3 | 5
  Second degree relative | 2 | 3 | 5
  Third degree relative or further removed | 0 | 1 | 1
Autoantibodies Positive [Count of Participants; unit: Participants]
  Anti-GAD65 harmonized | 40 | 28 | 68
  Micro insulin | 20 | 11 | 31
  Anti-IA-2 harmonized | 27 | 24 | 51
  Islet Cell Cytoplasmic Autoantibodies (ICA) | 29 | 28 | 57
  Anti-ZnT8 | 32 | 24 | 56
Glycated hemoglobin level [Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin] | 5.2 [4.9 to 5.4] | 5.3 [5.1 to 5.4] | 5.2 [5.0 to 5.4]

OUTCOME MEASURES:

1. Primary Outcome: Rate of New Diabetes Per Year
Description: Rate at which criteria are met for diabetes onset as defined by the American Diabetes Association (ADA) based on glucose testing or the presence of unequivocal hyperglycemia with acute metabolic decompensation.
Time Frame: During follow-up, median 745 days, range 74 to 2683
Population: Relatives of patients with type 1 diabetes who did not have diabetes but were at high risk for development of clinical disease.
Measure: Number; unit: N diabetes per 100 participant years
Arm/Group | Teplizumab | Placebo Infusion
Number analyzed (Participants) | 44 | 32
N diabetes per 100 participant years | 43 | 72

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events categorized and graded via CTCAE.
Time Frame: Baseline Visit to Diagnosis of Type 1 Diabetes median 745 days, range 74 to 2683
Measure: Count of Participants; unit: Participants
Arm/Group | Teplizumab | Placebo Infusion
Number analyzed (Participants) | 44 | 32
Participants | 43 | 23

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for individual participants, beginning with the Baseline Visit and ending with the documented Diagnosis of Type 1 Diabetes (the primary study endpoint), median 745 days, range 74 to 2683.
Description: CTCAE
Arm/Group | Teplizumab | Placebo Infusion
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/32
Serious Adverse Events (participants affected / at risk) | 8/44 | 1/32
Other Adverse Events (participants affected / at risk) | 43/44 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teplizumab (N=44) | Placebo Infusion (N=32)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection - Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Obstruction, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Obstruction, GU (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teplizumab (N=44) | Placebo Infusion (N=32)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (4) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2) | 0 (0)
Alpha-Gal Allergy (Immune system disorders) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (3) | 0 (0)
Dental: periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (3) | 0 (0)
Flu-like syndrome (General disorders) | 2 (7) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 2 (6) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with Normal ANC (Infections and infestations) | 12 (34) | 4 (13)
Infection with unknown ANC (Infections and infestations) | 5 (9) | 1 (3)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (13) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 30 (73) | 2 (5)
Leukocytes (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Mood alteration (Nervous system disorders) | 2 (4) | 2 (6)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (2)
Cognitive Disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (2) | 1 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (5) | 1 (6)
Obstruction, GI (Gastrointestinal disorders) | 1 (3) | 0 (0)
Ocular surface disease (Eye disorders) | 2 (4) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 10 (13) | 4 (6)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2)
Pulmonary/Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13 (41) | 0 (0)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (3)
Weight gain (General disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Breast function/lactation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Cardiac Arrhythmia - Other (Specify in Event Details) (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dental: teeth (Gastrointestinal disorders) | 0 (0) | 2 (4)
Dental: teeth development (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 2 (3)
Eyelid dysfunction (Eye disorders) | 0 (0) | 1 (2)
Elevated Bilirubin (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (2)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Personality/behavioral (Nervous system disorders) | 0 (0) | 1 (1)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-06-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT01030861/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT01030861/SAP_001.pdf